CLINICAL TRIAL: NCT02054845
Title: BEWARE: Body Awareness Training in the trEatment of Wearing-off Related Anxiety in Patients With paRkinson's diseasE.
Acronym: BEWARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Parkinsonvereniging (Unknown)
Responsible Party: Principal Investigator, O.A. van den Heuvel, Psychiatrist, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CWO/13-05E
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Parkinsonism, Experimental; Parkinsonism, Treatment as Usual
Keywords: Body awareness therapy; Physical therapy
MeSH Terms: conditions — Parkinsonian Disorders | interventions — Physical Therapy Modalities; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Body awareness therapy (Experimental): The experimental treatment: BEWARE
  Interventions: Behavioral: Body awareness therapy
- Treatment as Usual (Active Comparator): The new treatment is compared to this arm: Physical therapy
  Interventions: Other: Physical therapy

INTERVENTIONS:
Behavioral: Body awareness therapy — Experimental condition: BEWARE training group The physical and psychosocial elements of the training sessions will be complementary: psychological techniques are used to induce and endure wearing-off and physical techniques are used to improve body awareness to cope with the off-periods.
  Specifically the following techniques will be applied:
  1. Body scan
  2. Psychoeducation
  3. Acceptance Commitment Therapy / Mindfulness skills (sustained attention, concentration, non-reactivity, nonjudging of experience)
  4. Body Awareness Training
  5. Exposure training (imaginary exposure to induce response fluctuations)
  6. Training in cueing techniques to overcome problems with initiation and freezing
  7. Visual Feedback training
  8. Relaxation techniques
  Other Names: BEWARE
  Arms: Body awareness therapy
Other: Physical therapy — Control condition: Treatment as Usual The control group will receive treatment as usual based on the current guidelines for physical therapy in patients with Parkinson's Disease, with the same training schedule of 2x per week for 1,5 hours during 6 weeks. Group treatment will contain exercises for balance, walking, posture, transfers, arm/hand dexterity, strength, flexibility, relaxation and physical condition.
  Other Names: Treatment as usual
  Arms: Treatment as Usual

SUMMARY:
Approximately 60% of the patients with Parkinson's Disease (PD) that receive Levodopa therapy eventually develop response fluctuations in motor symptoms, such as rigidity, freezing and akinesia. Patients experience an 'off'-period just before the next dose of dopaminergic medication is needed, called the 'wearing-off'-phenomena. Wearing-off is also accompanied by non-motor symptoms such as depression, anxiety, pain and thinking disability. Together, these motor and non-motor symptoms have a major impact on the quality of life of patients and their partner or caregiver.

Patients with wearing-off often experience severe anxiety and panic symptoms that are incongruent with the severity of the motor symptoms during an 'off' period. These symptoms include stress, dizziness, pounding/racing of the heart, dyspnoea and hyperventilation. This type of anxiety is called wearing-off related anxiety (WRA) and might be a consequence of the hypersensitivity towards somatic manifestations and effects of a wearing-off period. This bodily misperception can have major consequences for the patient's feelings and behaviour. The experienced anxiety is often not consciously linked to the wearing-off and is therefore not well recognized by neurologists.

Treatment as usual in response fluctuations is physiotherapy, consisting of physical exercises for mobility problems, freezing, dyskinesias, etc. This kind of training hardly touches upon the mental aspects and the role of anxiety as integral element of the response fluctuations. Cognitive behaviour therapy (CBT, including exposure in vivo) is sometimes used to treat WRA, but seems to have unsatisfactory results since the changed body awareness is not sufficiently addressed. Also, the methods used in cognitive therapies focus on the elimination of WRA which is often not realistic since wearing-off symptoms will remain or even increase during disease progression. As of yet, there are no known alternative intervention options. This study focuses on a new intervention by integrating elements from physiotherapy, mindfulness, CBT (mainly exposure), Acceptance and Commitment Therapy (ACT) and psycho-education.

Objective: The current proposal aims at investigating the effect of a multidisciplinary non-verbal intervention on the awareness and modulation of WRA to improve self-efficacy, mobility, mood, and quality of life as compared to usual care.

Study design: Randomized controlled clinical trial.

Study population: Thirty-six PD patients who experience WRA.

Intervention: Patients with PD are randomly allocated into one of two groups (n= 18 each). One group receives the experimental 'body-awareness therapy', while the second group receives regular group-physiotherapy (treatment as usual). Both interventions will take 6 weeks in which 2 sessions per week with a duration of 1,5 hour will be performed.

Main study parameters/endpoints: The General Self-Efficacy Scale is the primary outcome measure and will be assessed prior to, directly after and 18 weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's Disease
* Experiencing Wearing-off
* Experiencing anxiety (BAI > 27)

Exclusion Criteria:

* Dementia (MMSE < 22)
* Other neurologic, orthopedic, cardiopulmonary problems that may interfere with participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy | Change from baseline in self-efficacy at 6 weeks
  how the patients can live their lives without being controlled by their disease, measured with the General Self Efficacy Scale
Self-efficacy | Change from baseline in self-efficacy at 18 weeks
  how the patients can live their lives without being controlled by their disease, measured with the General Self Efficacy Scale

SECONDARY OUTCOMES:
Anxiety | Change from baseline in anxiety at 6 weeks
  measured with the Beck Anxiety Inventory
Depression | Change from baseline in depression at 6 weeks
  measured with the Beck Depression Inventory
Balance performance | Change from baseline in balance performance at 6 weeks
  measured with the One Leg Stance test
comfortable walking speed | Change from baseline in walking speed at 6 weeks
  measured with the 10 Meter Walk Test
Quality of life | Change from baseline in quality of life at 6 weeks
  measured with the Parkinson's Disease Questionnaire - 39
Wearing-off symptoms | Change from baseline in wearing-off symptoms at 6 weeks
  Assessing wearing-off related symptoms with the Wearing-off Questionnaire - 19
Activities of Daily Living independence | Change from baseline in independence at 6 weeks
  measured with the Nottingham Extended Activities of Daily Living index
Freezing of Gait | Change from baseline in freezing of gait at 6 weeks
  To asses an important symptom of Parkinson's disease, we included the Freezing of Gait Questionnaire
Anxiety | Change from baseline in anxiety at 18 weeks
  measured with the Beck Anxiety Inventory
Depression | Change from baseline in depression at 18 weeks
  measured with the Beck Depression Inventory
Balance performance | Change from baseline in balance performance at 18 weeks
  measured with the One Leg Stance Test
Comfortable walking speed | Change from baseline in walking speed at 18 weeks
  measured with the 10 Meter Walk Test
Quality of Life | Change from baseline in quality of life at 18 weeks
  measured with the Parkinson's Disease Questionnaire - 39
Wearing-off symptoms | Change from baseline in anxiety at 6 weeks
  assessing wearing-off related symptoms with the Wearing-Off Questionnaire - 19
Activities of Daily Living independence | Change from baseline in independence at 18 weeks
  measured with the Nottingham Extended Activities of Daily Living index
Freezing of gait | Change from baseline in freezing of gait at 18 weeks
  to assess an important symptom of Parkinson's Disease, as measured by the freezing of gait questionnaire

OTHER OUTCOMES:
Mental state | baseline
  To decide whether patients have to be excluded from the study, cognitive ability is measured with the Mini Mental State Examination (MMSE)

CONTACTS AND LOCATIONS:
Overall Officials: O A van den Heuvel, psychiatrist, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Ghielen I, van Wegen EEH, Rutten S, de Goede CJT, Houniet-de Gier M, Collette EH, Burgers-Bots IAL, Twisk JWR, Kwakkel G, Vermunt K, van Vliet B, Berendse HW, van den Heuvel OA. Body awareness training in the treatment of wearing-off related anxiety in patients with Parkinson's disease: Results from a pilot randomized controlled trial. J Psychosom Res. 2017 Dec;103:1-8. doi: 10.1016/j.jpsychores.2017.09.008. Epub 2017 Sep 21. PMID 29167034
- [Derived] Ghielen I, van den Heuvel OA, de Goede CJ, Houniet-de Gier M, Collette EH, Burgers-Bots IA, Rutten S, Kwakkel G, Vermunt K, van Vliet B, Berendse HW, van Wegen EE. BEWARE: Body awareness training in the treatment of wearing-off related anxiety in patients with Parkinson's disease: study protocol for a randomized controlled trial. Trials. 2015 Jun 23;16:283. doi: 10.1186/s13063-015-0804-0. PMID 26101038
- See also: information on the BEWARE study — http://www.parkinson-beware.nl